CLINICAL TRIAL: NCT04700813
Title: Research Study for Rare Pathogenic Mutations Causing Type 2 Diabetes and Complications
Acronym: PreciDiag
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Collaborators: EGID, Lille (Unknown)
Responsible Party: Principal Investigator, Nicolas PAQUOT, Professor, University of Liege
Other Study IDs: 2019-166; B707201940651 (Other: numéro belge)
Record Dates: First submitted 2020-12-24; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — * 1 × 5mL of blood on EDTA for DNA extraction,
  * 4 × 5 mL of blood in a dry tube for the constitution of a serum bank,
  * 2 × 5 mL of blood on EDTA for the preservation of the plasma for the subsequent performance of additional analyzes as part of a positive genetic diagnosis.
  Au total : 35 mL de sang seront prélevés.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: search for rare pathogenic mutations — search for rare pathogenic mutations causing diabetes type 2

SUMMARY:
Single-center trial The goal is to better understand the various genetic mutations encountered in cases of type 2 diabetes as well as their frequency of occurrence in the population.

Such analyzes also make it possible to develop personalized medicine and to be able to prevent the associated risks.

The aim of this work is also to demonstrate the value of a systematic genetic diagnosis of patients with DMT2 in order to improve their clinical management.

Taking a blood sample, which will consist of the single sample from the entire study (1 single visit, combined with a follow-up visit to the patient's usual diabetist).

Participation in this study would make it possible to diagnose rare pathogenic mutations in type 2 diabetes and therefore to be able to adapt the treatment in a specific and personal way depending on the presence or not of the mutations and also to prevent the appearance of other pathologies.

DETAILED DESCRIPTION:
Procedure and methodology: during a follow-up visit to their usual diabetist (at CHU de Liège), we will send each potential volunteer, fulfilling the conditions for inclusion, an information and consent form relating to genetic analyzes. Participation in the protocol is voluntary, after detailed information and discussion with the patient. Once the participation agreement has been obtained, we will take a blood sample, which will be the only sample from the entire study.

All the tubes will be centrifuged, decanted, separated and frozen at -80 °C at the CHU de Liège for constitution of a serum bank on site, and of a DNA library at UMR8199.

For DNA extraction, samples will be sent at -80 ° C. DNA extraction will be automated (Autopure, Qiagen).

After DNA extraction, the genes involved in monogenic diabetes (Table 1) will be sequenced via Twist or NimbleGen capture in combination with Illumina sequencing (NovaSeq 6000), as recommended by Twist, NimbleGen and Illumina. The target will also include genes involved in the rare forms of metabolic diseases associated with diabetes: obesity, metabolic syndrome, familial hypercholesterolemia, kidney disease, cardiovascular disease and non-alcoholic fatty liver disease. This will help refine the patient's phenotypic understanding and improve their care.

Table 1. List of genes involved in monogenic diabetes

Gene ID NM ID ABCC8 NM_000352.4 APPL1 NM_012096.2 BLK NM_001715.2 CEL NM_001807.4 DNAJC3 NM_006260.4 DYRK1B NM_004714.2 EIF2AK3 NM_004836.5 FOXP3 NM_014009.3 GATA4 NM_002052.3 GATA6 NM_005257.5 GCK NM_000162.3 GLIS3 NM_152629.3 HNF1A NM_000545.5 HNF1B NM_000458.3 HNF4A NM_175914.4 IER3IP1 NM_016097.4 INS NM_000207.2 KCNJ11 NM_000525.3 KLF11 NM_003597.4 LRBA NM_6726.4 MAFA NM_201589.3 MNX1 NM_005515.3 MRAP2 NM_138409.3 NEUROD1 NM_002500.4 NEUROG3 NM_020999.3 NKX2-2 NM_002509.3 PAX4 NM_006193.2 PAX6 NM_000280.4 PCBD1 NM_000281.3 PDX1 NM_000209.3 PPP1R15B NM_032833.4 PTF1A NM_178161.2 RFX6 NM_173560.3 SLC19A2 NM_006996.2 SLC2A2 NM_000340.1 STAT3 NM_139276.2 TRMT10A NM_152292.4 WFS1 NM_006005.3 ZFP57 NM_001109809.2

Following sequencing, mutations will be detected and annotated according to the bioinformatics protocol implemented and optimized in UMR8199 since 2009.

Clinical and medical data will also be collected: weight, height, blood pressure, drug treatment, medical and surgical history as well as any other important medical information concerning the subject of the project. Data concerning the patient's ethnic origin will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2

Criteria exclusion:

* Refusal of participation
* Type 1 diabetic
* Presence of auto-antibodies directed against the β cells of the pancreas (insulin-secreting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients monitored for this pathology at the study site academic hospital of Liège
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
pathogenic mutations causing type 2 diabetes | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marjorie Fadeur, Liège, Belgium